CLINICAL TRIAL: NCT07177183
Title: Low Serum Creatinine as a Predictor of Prolonged Mechanical Ventilation and Weaning Failure
Acronym: SECRET-VENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KreaTINKA-2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prolonged Mechanical Ventilation; Critical Illness
Keywords: Prolonged mechanical ventilation; Critical illness; Creatinine; Creatine supplementation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: The patients will be randomised into three study arms (active treatment, placebo and controls)
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (control group) (Active Comparator): Patients with normal baseline serum creatinine value will be enrolled in this group. The care provided to patients in this group will not differ from the usual care provided to other patients.
  Interventions: Other: No intervention
- Group 2 (intervention group) (Experimental): Patients with subnormal baseline serum creatinine value will be randomly assigned to group 2 or 3. One group will receive creatine as a dietary supplement and the other will receive placebo. Other care provided to subjects in these groups will not differ from the usual care.
  Interventions: Dietary Supplement: Dietary supplement creatine
- Group 3 (intervention group) (Experimental): Patients with subnormal baseline serum creatinine value will be randomly assigned to group 2 or 3. One group will receive creatine as a dietary supplement and the other will receive placebo. Other care provided to subjects in these groups will not differ from the usual care.
  Interventions: Dietary Supplement: Dietary supplement - placebo

INTERVENTIONS:
Dietary Supplement: Dietary supplement creatine — Dietary supplement creatine. The dosage of creatine will be as follows: for the first 7 days after enrolment, the daily dose will be 2x5g. From days 8 to 21, the daily dose will be 1x5g. The substance will be administered orally or through a nasogastric tube.
  Arms: Group 2 (intervention group)
Dietary Supplement: Dietary supplement - placebo — Dietary supplement polydextrose as a placebo. The dosage of placebo will be as follows: for the first 7 days after enrolment, the daily dose will be 2x5g. From days 8 to 21, the daily dose will be 1x5g. The substance will be administered orally or through a nasogastric tube.
  Arms: Group 3 (intervention group)
Other: No intervention — Patients in Group 1 will serve as controls and will receive no intervention, only standard care.
  Arms: Group 1 (control group)

SUMMARY:
The main objective of the study is to determine whether a subnormal serum creatinine value upon admission to the Post-ICU Care Unit predicts the need for prolonged ventilatory support. A parallel objective of the study is to determine whether exogenous in-take of the dietary supplement creatine in patients with subnormal serum creatinine value is associated with a shortened duration of ventilatory support and improved patients outcome.

DETAILED DESCRIPTION:
More than 95% of serum creatinine comes from skeletal muscles, where it is formed by non-enzymatic degradation of creatine. Therefore, in patients with normal kidney function, the serum creatinine value closely correlates with muscle mass volume. It is well documented that critically ill patients lose almost 20% of their muscle mass volume during the first 10 days of their stay in the intensive care unit (ICU). At the same time, it is clear that it is from this group of "longer-stay" patients that those who need subsequent intensive care come. From the above, it can be assumed that in some patients admitted to the post-ICU care unit, the admission serum creatinine value may be subnormal due to muscle devastation caused during the stay in the ICU. This assumption was verified by analysing the admission creatinine values in a group of chronically ventilated adult patients admitted to the post-ICU care unit on CHRONICARE GROUP a.s. over five consecutive months. Of the total number of 264 patients, 123 (47%) patients had an admission serum creatinine value in the subnormal range.

Subnormal serum creatinine levels in patients admitted to the post-ICU care unit may have a number of causes, most of which are related to the patient's pre-existing illness, medical interventions in the ICU, or the critical illness itself. It may be related to chronic liver disease (suppressed creatine synthesis) or kidney disease (suppressed creatine synthesis). It may also be a falsely low serum creatinine level caused by fluid overload. Critical illness itself leads to sarcopenia, as a result of which the total amount of creatinine produced in the muscles decreases, and therefore the serum creatinine concentration. Unfortunately, the development of sarcopenia induced by critical illness cannot be influenced therapeutically. Similarly, mitochondrial dysfunction in muscle cells induced by critical illness cannot be influenced therapeutically. This abnormality leads to a decrease in Adenosine Triphosphate (ATP) production and therefore to a decrease in the formation of creatine phosphate, which is the main source for creatinine formation (the conversion of creatine phosphate to creatinine is 3 times faster than the conversion of creatine to creatinine). It is also possible that the subnormal value of serum creatinine is a consequence of an insufficient supply of creatine during nutritional support of critically ill patients in the ICU. Parenteral nutrition does not contain creatine at all, and enteral nutrition are mostly made from milk, which contains only minimal amounts of creatine. This fact creates an environment for the transformation of critically ill patients into the "position of vegetarians", who have demonstrably lower serum creatinine concentrations and also lower muscle strength than "omnivores".

A number of clinical studies have shown that low serum creatinine on admission are associated with higher mortality in patients admitted to the ICU. However, it is not known whether this finding also apply to patients admitted to the post-ICU care unit. Similarly, it is not known whether nutritional support enriched with creatine can improve the outcome of patients admitted to the ICU or to the post-ICU care units. Creatine is a food supplement with significant ergogenic potential and its beneficial effect in these patients is generally expected. The aim of the study is to contribute to clarifying the above-described uncertainties in the knowledge of this issue. The relationship between subnormal serum creatinine od admission and weaning from mechanical ventilation will be investigated through prospective observation, with the assumption that patients with subnormal creatinine levels will have a prolonged weaning compared to patients with normal creatinine values. The methodology of a prospective double-blind, placebo-controlled, randomized clinical trial will be used to investigate the benefit of supplementing nutritional support with creatine in a group of patients with subnormal creatinine value on admission. It is assumed that this procedure will be associated with a reduction in the need for ventilatory support and a better outcome compared to patients who will not receive creatine.

ELIGIBILITY:
Inclusion Criteria:

* Patients <18 years of age
* Patients admitted to post-ICU care units at Chronicare Group a.s. in the Czech Republic within 12 months

Exclusion Criteria:

* Patients who are unlikely to be weaned from ventilatory support.
* Patients in palliative care or with a survival probability of <3 months
* Patients with advanced malignancy
* Patients with a history of chronic kidney disease
* Patients with a history of chronic liver disease
* Patients with supranormal serum creatinine on admission to the post-ICU care unit
* Patients who refused to sign the Informed Consent with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free hours | 21 days
  The primary endpoint of the study will be the "ventilator-free hours", i.e. the total number of hours that the patient was without ventilator support

SECONDARY OUTCOMES:
Incidence of newly recorded infections | 21 days
  Secondary endpoints of the study will also include monitoring the incidence of newly recorded infections, assessing the level of respiratory effort with the use of a cough assist. The level of respiratory strength when using a cough assist will be assessed by measur-ing "Peak Cough Flow" directly on the device used. This will be assessed on study days 1, 7, 14, and 21 after enrolment. A newly recorded infection will be considered a situation where it was necessary to start a new antibiotic treatment or a situation where it was necessary to escalate an al-ready ongoing antibiotic treatment. The frequency of occurrence of these situations will be assessed daily over a 21-day period.
Changes in self-sufficiency | 21 days
  Changes in self-sufficiency will be assessed using the Barthel scale.
Changes in cognitive status | 21 days
  Changes in cognitive status will be assessed using the "ChroniCare Cognitive Orientation Tool (CC-COT)", a non-standardized tool for the assessment of cognition in patients with limited verbal and non-verbal communication. The tool is a modification of the Mini-Cog test that has been adapted for the conditions of the post-ICU care in patients with tracheostomy, ventilator support, and limited verbal and non-verbal communication.
Changes in muscle strength | 21 days
  Changes in muscle strength will be assessed using a hand-held dynamometer.
Creatine tolerance | 21 days
  To assess creatine tolerance, the incidence of gastrointestinal discomfort (bloating or diarrhoea) will be monitored daily for 21 days. The incidence of creatinine and cystatin C elevations into the supranormal range will also be monitored on days 7, 14, and 21 after study enrolment.

OTHER OUTCOMES:
28-day mortality | 28 days
  28-day mortality will be monitored as a tertiary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Kula, MD, CSc, Study Chair — University Hospital Ostrava
Locations (2):
- Czechia (2):
  - Chronicare Mund s.r.o., Brno
  - Chronicare s.r.o., Milovice

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan to share individual participant data with other researchers. The data may be provided upon reasonable request.

REFERENCES:
- [Background] Williamson L, New D. How the use of creatine supplements can elevate serum creatinine in the absence of underlying kidney pathology. BMJ Case Rep. 2014 Sep 19;2014:bcr2014204754. doi: 10.1136/bcr-2014-204754. PMID 25239988
- [Background] Groeneveld GJ, Beijer C, Veldink JH, Kalmijn S, Wokke JH, van den Berg LH. Few adverse effects of long-term creatine supplementation in a placebo-controlled trial. Int J Sports Med. 2005 May;26(4):307-13. doi: 10.1055/s-2004-817917. PMID 15795816
- [Background] Gala K, Desai V, Liu N, Omer EM, McClave SA. How to Increase Muscle Mass in Critically Ill Patients: Lessons Learned from Athletes and Bodybuilders. Curr Nutr Rep. 2020 Dec;9(4):369-380. doi: 10.1007/s13668-020-00334-0. PMID 33098051
- [Background] Thongprayoon C, Cheungpasitporn W, Kittanamongkolchai W, Harrison AM, Kashani K. Prognostic Importance of Low Admission Serum Creatinine Concentration for Mortality in Hospitalized Patients. Am J Med. 2017 May;130(5):545-554.e1. doi: 10.1016/j.amjmed.2016.11.020. Epub 2016 Dec 18. PMID 27998681
- [Background] Thongprayoon C, Cheungpasitporn W, Kashani K. Serum creatinine level, a surrogate of muscle mass, predicts mortality in critically ill patients. J Thorac Dis. 2016 May;8(5):E305-11. doi: 10.21037/jtd.2016.03.62. PMID 27162688
- [Background] Sahin Tutak A, Aydin H, Findikli HA. Prognostic significance of low basal serum creatinine levels in internal intensive care unit patients. Eur Rev Med Pharmacol Sci. 2023 Jan;27(2):592-600. doi: 10.26355/eurrev_202301_31060. PMID 36734702
- [Background] Cartin-Ceba R, Afessa B, Gajic O. Low baseline serum creatinine concentration predicts mortality in critically ill patients independent of body mass index. Crit Care Med. 2007 Oct;35(10):2420-3. doi: 10.1097/01.ccm.0000281856.78526.f4. PMID 17948336
- [Background] Bartholomae E, Knurick J, Johnston CS. Serum creatinine as an indicator of lean body mass in vegetarians and omnivores. Front Nutr. 2022 Sep 16;9:996541. doi: 10.3389/fnut.2022.996541. eCollection 2022. PMID 36185683
- [Background] Fredriksson K, Hammarqvist F, Strigard K, Hultenby K, Ljungqvist O, Wernerman J, Rooyackers O. Derangements in mitochondrial metabolism in intercostal and leg muscle of critically ill patients with sepsis-induced multiple organ failure. Am J Physiol Endocrinol Metab. 2006 Nov;291(5):E1044-50. doi: 10.1152/ajpendo.00218.2006. Epub 2006 Jun 27. PMID 16803854
- [Background] Klawitter F, Ehler J, Bajorat R, Patejdl R. Mitochondrial Dysfunction in Intensive Care Unit-Acquired Weakness and Critical Illness Myopathy: A Narrative Review. Int J Mol Sci. 2023 Mar 14;24(6):5516. doi: 10.3390/ijms24065516. PMID 36982590
- [Background] Jiroutkova K, Krajcova A, Ziak J, Fric M, Waldauf P, Dzupa V, Gojda J, Nemcova-Furstova V, Kovar J, Elkalaf M, Trnka J, Duska F. Mitochondrial function in skeletal muscle of patients with protracted critical illness and ICU-acquired weakness. Crit Care. 2015 Dec 24;19:448. doi: 10.1186/s13054-015-1160-x. PMID 26699134
- [Background] Yamamoto N, Tojo K, Mihara T, Maeda R, Sugiura Y, Goto T. Creatinine production rate is an integrative indicator to monitor muscle status in critically ill patients. Crit Care. 2025 Jan 14;29(1):23. doi: 10.1186/s13054-024-05222-5. PMID 39810218
- [Background] Lieu C, Anderson R. Serum creatinine: why lower may not be better. Crit Care Med. 2007 Oct;35(10):2458-9. doi: 10.1097/01.CCM.0000284738.81354.FC. No abstract available. PMID 17885392
- [Background] Heimburger O, Stenvinkel P, Barany P. The enigma of decreased creatinine generation in acute kidney injury. Nephrol Dial Transplant. 2012 Nov;27(11):3973-4. doi: 10.1093/ndt/gfs459. No abstract available. PMID 23144066
- [Background] Assy N, Kayal M, Mejirisky Y, Gorenberg M, Hussein O, Schlesinger S. The changes in renal function after a single dose of intravenous furosemide in patients with compensated liver cirrhosis. BMC Gastroenterol. 2006 Nov 29;6:39. doi: 10.1186/1471-230X-6-39. PMID 17134488
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Kim SW, Jung HW, Kim CH, Kim KI, Chin HJ, Lee H. A New Equation to Estimate Muscle Mass from Creatinine and Cystatin C. PLoS One. 2016 Feb 5;11(2):e0148495. doi: 10.1371/journal.pone.0148495. eCollection 2016. PMID 26849842